CLINICAL TRIAL: NCT03541031
Title: Micronutrients as Adjunctive Treatment for Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Maine Medical Center (Other)
Responsible Party: Principal Investigator, Lewis Mehl-Madrona, MD, Principal Investigator, Eastern Maine Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 17-1-M-354
Record Dates: First submitted 2017-12-12; First posted 2018-05-30 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Micronutrients; Fish Oils; Olive Oil; Safflower Oil

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized clinical trial that will assign 120 stable adult outpatients with bipolar disorder, type I or II (DSM-V criteria) to supplementation with a 36-ingredient vitamin/mineral mix (Micronutrient) and an omega-3 fatty acid supplement (Fish oil) (N=72) or to matched double placebo (N=48) in a 3:2 ratio for a year.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only one individual (unblind coordinator) will know which patients are receiving placebo and which are receiving active micronutrients. She will have no contact with the subjects. All research and clinical staff and all patients will be blinded to what they are actually receiving. The unblind coordinator has verified that the placebos appear identical in appearance to the active micronutrients. The placebos have been manufactured by the same companies that make the actual micronutrients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Micronutrient & Fish oil (Experimental): Fish oil capsule by mouth 3 capsules daily, remaining constant throughout the study and Micronutrient capsule by mouth beginning with a fixed schedule of 2 capsules twice daily and increasing monthly by 2 capsules twice daily up to a maximum of 16 capsules/day.
  Interventions: Dietary Supplement: Micronutrient & Fish oil
- Olive oil & Safflower oil (Placebo Comparator): Safflower oil capsule by mouth 3 capsules daily, remaining constant throughout the study and Olive oil capsule by mouth beginning with a fixed schedule of 2 capsules twice daily and increasing monthly by 2 capsules twice daily up to a maximum of 16 capsules/day.
  Interventions: Dietary Supplement: Olive oil & Safflower oil

INTERVENTIONS:
Dietary Supplement: Micronutrient & Fish oil — Capsule containing a 36-ingredient micronutrient formula (EMPowerplus™) which has been widely researched for its usefulness in several psychiatric conditions. The second product is a capsule containing Fish oil (Wiley's Finest™ Wild Alaskan Fish Oil Peak EPA; 700 mg EPA plus DHA per capsule).
  Other Names: EMPowerplus™ & Peak EPA
  Arms: Micronutrient & Fish oil
Dietary Supplement: Olive oil & Safflower oil — Olive oil capsule manufactured to mimic Micronutrient and safflower oil capsule manufactured to mimic Fish oil
  Arms: Olive oil & Safflower oil

SUMMARY:
The purpose of the trial is to determine whether a 36-ingredient Micronutrient supplement (primarily vitamins and minerals) and Fish oil (omega-3 fatty acid) supplement improves nutritional status and allows lower doses of conventional medications to be effective for bipolar disorder with fewer side effects, when studied under randomized and fully blinded conditions and compared to a placebo. All participants must live in the vicinity of Bangor, Maine.

DETAILED DESCRIPTION:
Bipolar disorder is a common neuropsychiatric illness with high rates of morbidity and mortality. Despite available medications to treat bipolar disorder, recurrence rates are high. Bipolar disorder is conventionally treated with typical or antipsychotic medications are well described and include the increased risk of acute kidney injury, cataracts, decreased cognitive function, increased risk for myocardial infarction and stroke, metabolic syndrome and type 2 diabetes mellitus, and dyslipidemia. Related to this, mortality rates are elevated among people with bipolar disorder compared to the general population. Men with the diagnosis of bipolar disorder live, on average 13.6 years less than the general population, and for women, 12.1 years less.

This RCT (randomized clinical trial) compares a 36-ingredient Micronutrient supplement and Fish oil supplement to matched double placebo in patients randomized to receive one or the other for 52 weeks. One hundred twenty (120) patients are randomized in a 3:2 ratio to Micronutrient + Fish oil or to placebo, respectively. All patients are stably medicated adult outpatients with bipolar disorder (type I or type II). Medical supervision is provided with monthly appointments. At the end of the 52 weeks, all participants will be offered the opportunity of entering a 52-week open-label extension. The primary hypothesis is that active supplementation will allow significantly more reduction of conventional medication than placebo will, without a significant increase in symptoms and with significantly fewer side effects/adverse events.

The objective of this study is to assess the efficacy of Micronutrient supplement + Fish oil compared with placebo in stably medicated adults with bipolar disorder I and II, in improving nutritional status, allowing conventional medication to be effective at lower doses and with fewer side effects at the end of 52 weeks of therapy as assessed under randomized and fully blinded conditions. The primary outcome measure is a composite z-score for side effects, calculated from three separate z-scores that measure medication dosage, illness intensity (Clinical Global Impression score), and adverse side effects (UKU Side Effect score). Secondary outcomes include

* Symptom severity using the Positive and Negative Symptom Scale (PANSS)
* Mania symptoms using the Young Mania Rating Scale (YMRS)
* Anxiety symptoms using the Hamilton Anxiety scale (Ham-A)
* Depression symptoms using the Montgomery-Asberg Depression Rating Scale (MADRS)
* Quality of life, patient-reported using My Medical Outcome Profile version 2 (MYMOP-2)
* Nutritional status using the Mini Nutritional Assessment scale (MNA)
* Functionality, patient-reported using the 24-item Behavior and Symptom Identification Scale (BASIS-24)
* Vital signs (waist circumference, body mass index, blood pressure, heart rate, and respirations)

Treatment-emergent adverse events are documented at each appointment using the Adverse Event Log. Participants are screened and their suitability for the trial confirmed at the first visit. If suitability is confirmed, informed consent is obtained and they enter the randomized phase. Participants are seen monthly for 12 months, at which time (1) their medication is optimized (graded reduction in dose by 10% per month, upwards if symptoms are above the acceptable level and downwards if an acceptable level of symptom relief has been achieved); (2) symptoms and side effects are recorded; and (3) questionnaires are administered.

ELIGIBILITY:
Inclusion Criteria:

Individuals enrolled will be adult outpatients with a diagnosis of bipolar disorder I or II, receiving care at the Family Medicine Center & Residency Program of Eastern Maine Medical Center in Bangor, Maine. Participants must be able to complete questionnaires and examinations and comply with protocols.

Exclusion Criteria:

Participants will be excluded from the study for any of the following reasons:

1. Evidence of untreated or unstable thyroid disease (until it is treated and stabilized).
2. Known abnormality of mineral metabolism (e.g., Wilson's disease) until stabilized.
3. Unable to speak English
4. Any hypervitaminosis syndrome
5. Acute suicidality (until stabilized).

Participation in the study will not alter the participants' clinical care except that they will be provided Micronutrients and Fish oil (or placebos for each) and will participate in a monthly evaluation of the effect of adding these Micronutrients. We will ask them what other supplements they are taking and will instruct them not to take supplements that contain any of the same ingredients that they will receive in the study so as to avoid exceeding the maximum dose allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Side Effects | Baseline and every month for 1 year
  A composite z-score calculated from three separate z-scores for: (1) medication dosage, measured in haloperidol equivalents, valproic acid equivalents, lithium dose, fluoxetine equivalents, or lorazepam equivalents; (2) Clinical Global Impression (CGI) score, a measure of schizophrenia symptoms and illness at the time of assessment, with scores ranging from 1 (not at all ill) to 7 (extremely ill); and (3) UKU Side Effect score, which rates 48 single items of adverse side effects, clustered into four subgroups (psychic, neurological, autonomic and other side effects), on a scale of 1 to 4.

SECONDARY OUTCOMES:
Changes in Symptom Severity | Baseline and every 3 months for 1 year
  Scores on the Positive and Negative Symptom Scale (PANSS): The PANSS is a medical scale used to measure symptom severity of patients with schizophrenia. Of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale. Each of the 30 items is accompanied by a specific definition as well as detailed anchoring criteria for all seven rating points. These seven points represent increasing levels of psychopathology and range from 1 (absent) to 7 (extreme). The scores for these scales are arrived at by summation of ratings across component items. A Composite Scale is scored by subtracting the negative score from the positive score. This yields a bipolar index that ranges from -42 to +42, which is a difference score reflecting the degree of predominance of one syndrome in relation to the other.
Changes in Mania Symptoms | Baseline and every 3 months for 1 year
  Scores on the Young Mania Rating Scale (YMRS): The YMRS consists of 11 items. Items 5, 6, 8, and 9 are rated on a scale from 0 (symptoms not present) to 8 (symptoms extremely severe). The remaining items are rated on a scale from 0 (symptoms not present) to 4 (symptoms extremely severe). Items 5, 6, 8, and 9 (irritability, speech, content and disruptive-aggressive behavior) are given twice the weight of the remaining seven in order to compensate for the poor condition of severely ill subjects.
Changes in Anxiety Symptoms | Baseline and every 3 months for 1 year
  Scores on the Hamilton Anxiety Scale (Ham-A): The Ham-A is a widely used interview measure designed to assess anxiety (Hamilton, 1969). It consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe). The Ham-A features both psychic and somatic anxiety subscales. The psychic subscale, which is comprised of items that address the more subjective cognitive and affective components of anxious experience (e.g., anxious mood, tension, fears, difficulty concentrating), is particularly useful in assessing the severity of anxiety. In contrast, the somatic subscale emphasizes features of anxiety that are somewhat less typical, including autonomic arousal, respiratory and cardiovascular symptoms.
Changes in Depression | Baseline and every 3 months for 1 year
  Scores on the Montgomery-Asberg Depression Rating Scale (MADRS): The MADRS (Montgomery & Asberg, 1979), one of the most frequently used and validated observer-rated depression scales, is a 10-item rating scale to assess the severity of depressive symptoms within the last 7 days. The 10 selected items are rated on a scale of 0-6 with anchors at 2-point intervals. The interviewer is encouraged to use his or her observations of the patient's mental status as an additional source of information.
Changes in Quality of Life (patient-reported) | Baseline and every month for 1 year
  Scores on the My Medical Outcome Profile version 2 (MYMOP-2): The Health Services Research Collaboration of the UK's Medical Research Council has put together an individualized self-report measure called the MYMOP (Measure Yourself Medical Outcome Profile). The patient selects 2 symptoms to monitor --- things that matter to him/her. They also monitor 2 other things: an activity, and general sense of wellbeing. Medications are monitored as well.
  The quality of life between groups will be assessed.
Changes in Nutritional Status | Baseline and every 4 months for 1 year
  Scores on the Mini Nutritional Assessment (MNA) Scale: The MNA, at baseline and at four month intervals, is a validated nutrition screening and assessment tool that can identify patients at risk of malnutrition. The MNA was developed nearly 20 years ago and is the most well validated nutrition screening tool (Vellas, et al., 2006). There is a long and a short form. We will use the long form to more readily distinguish among levels of nutrition as opposed to just identifying those who are malnourished. It has been well validated in multiple populations and clinical settings (Bastiaanse, et al., 2011).
Changes in Functionality (patient-reported) | Baseline and every 3 months for 1 year
  Scores on the Behavior and Symptom Identification Scale (BASIS-24): The BASIS-24 is a 24 item patient self-report questionnaire designed to assess treatment outcomes by measuring symptoms and functional difficulties experienced by patients seeking mental health services. Items are scored using a weighted average algorithm that gives an overall score and scores for six subscales: Depression and Functioning, Relationships, Self-Harm, Emotional Liability, Psychosis, and Substance Abuse. All items are answered on a 5 point scale.
  The degree to which the illness restricts activities will be assessed between groups.
Changes in Waist Circumference | Baseline and every 4 months for 1 year
  Waist circumference (WC) is measured in cm.
Changes in Basal Metabolic Index | Baseline and every 4 months for 1 year
  Basal Metabolic Index (BMI) is measured in kg/m2.
Changes in Blood Pressure | Baseline and every 4 months for 1 year
  Blood pressure (BP) is measured in mmHg.
Changes in Heart Rate | Baseline and every 4 months for 1 year
  Heart rate is measured in beats per minute.
Changes in Respirations | Baseline and every 4 months for 1 year
  Respiration is measured in breaths per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Mehl-Madrona, MD, PhD, Principal Investigator — Eastern Maine Medical Center
Locations (1):
- Eastern Maine Medical Center, Bangor, Maine, United States

IPD SHARING:
Plan to Share IPD: Undecided